CLINICAL TRIAL: NCT06181565
Title: The Impact of Pericardial Closure on the Grafts, in the Context of Coronary Artery Bypass Grafting
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1342021/CHUSTE
Record Dates: First submitted 2023-11-23; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-11

CONDITIONS: Bypass Graft Stenosis
Keywords: Cardiac surgery; pericardial closure; grafts; bypass; aortocoronary bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who will have isolated aortocoronary bypass grafting surgery: Patients who will have isolated aortocoronary bypass grafting surgery will be included.
  The Medistim machine will be use before and after pericardial closure. Datas will be collected and analysis.
  Interventions: Other: Datas of Medistim machine

INTERVENTIONS:
Other: Datas of Medistim machine — Datas will be collected by Medistim machine before and after pericardial closure: Flow through the grafts, Resistance on grafts, Pulsatility of the grafts, Systolic and diastolic curves before and after pericardial closure
  Other Names: Medistim machine

SUMMARY:
Once the pericardium is closed, there is no information on the hemodynamics of the grafts after coronary artery bypass grafting. This would be the reason for different opinions on pericardial closure: some teams do not close the pericardium and others close it.

In the department Cardiovascular Surgery of the University Hospital of Saint-Etienne, the Medistim machine is used in routine and the hemodynamic properties of the grafts are recorded immediately after the bypass surgery, before the closure of the pericardium.

DETAILED DESCRIPTION:
The aim of the study is to have hemodynamic information immediately after the closure of the pericardium using the Medistim machine. The prospective study will be conducted on 50 patients, who will be selected consecutively without randomization. The inclusion and exclusion criteria are determined.

ELIGIBILITY:
Inclusion Criteria:

* All patients who will have isolated aortocoronary bypass grafting surgery

Exclusion Criteria:

* History of thoracic trauma
* Severe cyphosis
* Severe thoracic deformity (Pectus excavatum)
* Pericardial disease
* History of radiotherapy
* Severe pulmonary disease (emphysema)
* Right heart failure
* Redo surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who will have isolated aortocoronary bypass grafting surgery will be included.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Flow through the grafts | Minute : 1, 15
  Datas will be collected by Medistim machine.

SECONDARY OUTCOMES:
Resistance on grafts | Minute : 1, 15
  Datas will be collected by Medistim machine.
Pulsatility of the grafts | Minute : 1, 15
  Datas will be collected by Medistim machine.
Systolic curves | Minute : 1, 15
  Datas will be collected by Medistim machine.
Diastolic curves | Minute : 1, 15
  Datas will be collected by Medistim machine.

CONTACTS AND LOCATIONS:
Overall Officials: Andranik PETROSYAN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No